CLINICAL TRIAL: NCT06477406
Title: Evaluating the Impact of a Novel Cannabinoid Product for Endometriosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Massachusetts Life Sciences Center (Unknown)
Responsible Party: Principal Investigator, Staci Gruber, Ph.D., Director, Marijuana Investigations for Neuroscientific Discovery (MIND); Director, Cognitive and Clinical Neuroimaging Core (CCNC), Mclean Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024P001549
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-CBD Sublingual Product (Experimental): A custom-formulated, hemp-derived, full-spectrum high-CBD sublingual solution; 0.75mL of solution will be self-administered three times daily (TID) for the duration of the CBD phase.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Placebo solution (0.75mL) will be self-administered TID for the duration of the placebo phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Custom formulation of a hemp-derived sublingual solution that is high in CBD and includes other cannabinoids and terpenes.
  Arms: High-CBD Sublingual Product
Drug: Placebo — An active placebo containing supplemental terpenes matched to the high-CBD product.
  Arms: Placebo

SUMMARY:
Despite the proliferation of cannabis and cannabinoid products in recent years, little research has been done to determine the impact of these products on womens health conditions, including endometriosis. This study is designed to assess the impact of a custom-formulated, hemp-derived, full-spectrum, high-CBD product vs. placebo on clinical symptoms and biomarkers over the course of 12 weeks of treatment in patients with endometriosis. This project will provide information that does not currently exist on the potential efficacy of a cannabinoid-based sublingual product for endometriosis.

DETAILED DESCRIPTION:
Despite recent increases in both medical and recreational cannabis use in the United States and globally, little research has been conducted to determine the potential applications for womens health. Endometriosis impacts approximately 10% of women of reproductive age, an estimated 176 million individuals, and is characterized by endometrial cells growing outside of the uterus, resulting in severe pain, chronic inflammation, gastrointestinal symptoms, infertility, and often, depression and anxiety (WHO, 2023). Existing treatment options are often limited in efficacy and may result in a variety of negative side effects. Previous research has indicated that cannabinoids including cannabidiol (CBD), delta-9 tetrahydrocannabinol (THC), and a number of other cannabinoids may hold potential for treating the symptoms of endometriosis, especially the chronic pain associated with the condition.

This study is a double-blind crossover clinical trial of a high-CBD product compared to placebo over a total of 12 weeks of treatment in patients with endometriosis. Participants will complete 7 visits over 12 weeks; 4 visits will be conducted in-person at McLean Hospital in Belmont, MA, and 3 visits will be conducted remotely. Visits consist of clinical ratings, assessments of conventional medication use, quality of life measures, and providing saliva, urine, and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent
2. Sex assigned female at birth
3. Subject is 21 or older
4. Subject is fluent in English
5. Subject endorses at least moderate levels of pain at the baseline visit
6. Subject endorses having endometriosis

Exclusion Criteria:

1. Non-fluent English speakers
2. Endorsement of current substance use disorder, psychotic disorder, or an eating disorder
3. Currently uses cannabis or cannabinoid products regularly
4. Patients will be excluded if they have a positive urine pregnancy test, are trying to become pregnant, or are currently breastfeeding
5. Presence of a serious or unstable medical illness, including liver, kidney, or cardiovascular disease (hyper/hypotension, cardiac disorders), or neurological disorder (including seizure disorder)
6. Neuropathic pain or cancer-related pain
7. Disclosure of a genetic polymorphism affecting CYP2C9 function

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 weeks
  The VAS is a commonly used pain scale where patients draw a line to indicate their pain level on a 100 millimeter long line anchored by two verbal descriptors for symptom extremes (e.g. "no pain" to "worst imaginable pain"). The VAS will be used to describe different types of endometriosis-related pain (dysmenorrhea (pain during menstruation), dyspareunia (pain during or after intercourse), and non-menstrual chronic pelvic pain). Lower scores indicate less pain.

SECONDARY OUTCOMES:
Endometriosis Health Profile (EHP-30) | 12 weeks
  The EHP-30 is a well-validated self-report scale with 30 core items and 23 additional questions related to specific modules and areas of life often impacted by endometriosis symptoms. Lower scores indicate fewer symptoms.
VAS-IBS | 12 weeks
  The VAS-IBS queries bowel-related concerns. While initially developed for IBS patients, it is commonly used to assess gastrointestinal symptoms in endometriosis patients. Lower scores indicate fewer bowel symptoms.
Beck Anxiety Inventory (BAI) | 12 weeks
  The BAI is a 21 item-self-report measure that can be used to screen for anxiety. Each item on the BAI is rated on a scale of 0 to 3, and is descriptive of subjective, somatic, or panic-related symptoms of anxiety. Lower scores indicate fewer symptoms of anxiety.
Beck Depression Inventory (BDI) | 12 weeks
  The BDI is a 21 item-self-report measure that can be used to assess the severity of depression. Each item on the BDI relates to a symptom of depression and is rated by the subject using a 0-3 scale. Lower scores indicate fewer depressive symptoms.
Conventional Medication Use | 12 weeks
  Changes in conventional medication use will be assessed over the course of treatment with study product.
Inflammatory Biomarkers | 12 weeks
  Saliva samples will be used to quantify levels of common inflammatory markers (e.g. IL-1β, IL-6, IL-8, TNF-α). Lower levels of inflammatory markers indicate less systemic inflammation.
Circulating Endocannabinoid Concentrations | 12 weeks
  Plasma will be analyzed for circulating levels of endocannabinoids and related compounds (e.g., AEA, 2-AG, 2-OG, PEA, OEA).

CONTACTS AND LOCATIONS:
Overall Officials: Staci Gruber, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided